CLINICAL TRIAL: NCT02942628
Title: Vegetarian Diet in Patients With Ischemic Heart Disease: An Open-label, Randomized, Prospective Crossover Study
Brief Title: Vegetarian Diet in Patients With Ischemic Heart Disease
Acronym: VERDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Göteborg University (Other); Swedish University of Agricultural Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Regionorebrolan
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegetarian - Meat (Experimental): 4 weeks of vegetarian diet followed by 4 weeks of 'wash out' (no intervention) and 4 weeks of meat-containing diet
  Interventions: Other: Vegetarian diet followed by meat diet or vice versa
- Meat - Vegetarian (Active Comparator): 4 weeks of meat-containing diet followed by 4 weeks of 'wash out' (no intervention) and 4 weeks of vegetarian diet
  Interventions: Other: Vegetarian diet followed by meat diet or vice versa

INTERVENTIONS:
Other: Vegetarian diet followed by meat diet or vice versa — Half the patients will follow either a vegetarian diet for 6 weeks and the other half will adhere to or a meat-based diet for six weekd. This is followed by a 4 week period where patients eat their usual diet. Thereafter patients initially randomized to a vegetarian diet will follow a meat-based diet for six weeks while the patients initially randomized to meat will follow a vegetarian diet for six weeks.

SUMMARY:
Open label, 4 week randomized, cross-over study to compare the effect of a vegetarian diet to a conventional (meat containing) diet based on the Swedish average meat consumption on a range of parameters with prognostic importance for cardiovascular disease.The study will be conducted in patients diagnosed with ischemic heart disease. We hypothesize that patients will benefit from a vegetarian diet as assessed by multiple risk markers for this type of disease with a primary focus on changes in oxidized LDL cholesterol.

DETAILED DESCRIPTION:
Background

Cardiovascular disease is the leading cause of death globally. Ischemic heart disease (IHD) contributes the most to this statistic and since 1990 the global burden of IHD has increased. It is estimated that 50 000 Swedish patients are hospitalized every year due to IHD. The risk of developing IHD is to a large extent determined by the existence and state of several modifiable risk factors including dietary habits, smoking, hypertension, diabetes mellitus, hyperlipidemia, high apolipoprotein B/ apolipoprotein A1-ratio, abdominal obesity, physical inactivity, alcohol consumption and psychosocial factors. High levels of oxidative stress, oxidized LDL cholesterol and the microbial metabolite trimethylamine N-oxide TMAO have been suggested to be associated with development of IHD.

A plant-based (vegetarian) diet may provide cardiovascular health benefits through various mechanisms. Clinical studies suggest that a vegetarian diet has positive effects on low-density lipoprotein (LDL) cholesterol, oxidized LDL cholesterol, total cholesterol, triglycerides, apolipoprotein B, body mass index (BMI), inflammatory markers, blood pressure, arterial intima-media thickness, insulin sensitivity, glycated hemoglobin, (HbA1c) and fasting glucose levels. Through positive impacts on risk factors that a vegetarian diet is associated with a lowered incidence and mortality of IHD and an overall reduced mortality.

A weakness of several prior long-term controlled studies comparing vegetarian and meat-containing diets is the lack of well-defined control diets leading to study heterogeneity. For example, some of the subjects on meat-containing diets consume great quantities of red meat, others eat substantial amounts of processed meat products and some eat mostly white meat and fish complicating interpretation of outcome. In cross-sectional or observational cohort studies comparing long-term vegetarians to long-term omnivores, results may be influenced by other lifestyle choices besides the studied diet, such as smoking and exercise.Furthermore, the participants in many previous studies were often healthy volunteers and not patients with overt cardiovascular disease.

Purpose

The objective is to perform an open label, 4 week randomized, cross-over study to compare the effect of a vegetarian diet to a conventional (meat containing) diet based on the Swedish average meat consumption on a range of parameters with prognostic importance for cardiovascular disease: lipids, inflammation, oxidative stress, BMI, HbA1c, apolipoprotein B/apolipoprotein A1-ratio, gut microbiota, endothelial function and quality of life. The study will be conducted in patients diagnosed with STEMI (ST-segment elevation myocardial infarction), non-STEMI (non-ST-segment elevation myocardial infarction) or angina pectoris and treated by percutaneous coronary intervention (PCI).

Hypothesis

The study hypothesis is that patients diagnosed with IHD can benefit from a vegetarian diet as assessed by multiple risk markers for this type of disease with a primary focus on changes in oxidized LDL cholesterol.

Clinical relevance

During the last decades the global mortality from IHD has remained unchanged regardless of development of new invasive and pharmacological treatments. Despite the fact that the prevalence and mortality from IHD have decreased in this country since 1990 and that the decrease most likely is due to lifestyle changes, IHD remains the leading cause of death in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Stable ischemic heart disease and previous percutaneous coronary intervention (PCI.
* Under optimal medical treatment including aspirin and cholesterol lowering drugs (statins)

Exclusion Criteria:

* PCI treatment during the last 30 days
* Inability to provide informed consent
* Already following a vegetarian or a vegan diet
* Known vitamin B deficiency
* Known food allergy
* Previous obesity surgery or gastric bypass surgery
* Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in oxidative stress evaluated by oxidized LDL cholesterol changes | 4 weeks

SECONDARY OUTCOMES:
Changes in cardiovascular risk profile according to the Framingham Risk Score | 4 weeks
Changes in biomarkers of inflammation | 4 weeks
  Markers: hs-CRP (high sensitivity C-reactive protein), IL-6 (interleukin 6), TNF-α (tumor necrosis factor α), interferon gamma (IFN-γ).
Changes in biomarkers of lipid status | 4 weeks
  Markers: total cholesterol, LDL-cholesterol, TGA (triacylglycerides), apolipoprotein B, apolipoprotein A1, HDL cholesterol.
Changes in HbA1c | 4 weeks
Changes in TMAO levels in plasma | 4 weeks
  TMAO: trimethylamine N-oxide assessed by stable isotope dilution high-performance liquid chromatography.
Changes in gut microbiota | 4 weeks
  Assessment of: Bacteroides, Prevotella, Bacteroides-Prevotella, Bacteroides thetaiotaomicron, Clostridium clostridioforme and Faecalibacterium prausnitzii and 16S rRNA profiling and next-generation sequencing to analyze the gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Demir Djekic, MD, Principal Investigator — Region Örebro County
Locations (1):
- Regionorebrolan, Örebro, Sweden

REFERENCES:
- [Derived] Djekic D, Shi L, Brolin H, Carlsson F, Sarnqvist C, Savolainen O, Cao Y, Backhed F, Tremaroli V, Landberg R, Frobert O. Effects of a Vegetarian Diet on Cardiometabolic Risk Factors, Gut Microbiota, and Plasma Metabolome in Subjects With Ischemic Heart Disease: A Randomized, Crossover Study. J Am Heart Assoc. 2020 Sep 15;9(18):e016518. doi: 10.1161/JAHA.120.016518. Epub 2020 Sep 6. PMID 32893710